CLINICAL TRIAL: NCT05994651
Title: Evaluation of the Effect of Tidal Model on Distress, Self-Management and Psychological Well-Being in Individuals With Diabetes
Brief Title: The Effect of the Tidal Model in Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Ejdane Coskun, Lecturer, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Tidal Model
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Diabetic
Keywords: Diabetes disease; Psychiatric Nursing; Tidal Model; Psychological well-being; Distress; Self-Management
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tidal Model improvement model (Experimental): In order to provide individualized care to the individuals in the experimental group, initiatives will be implemented by starting individual interviews and in line with the goals of the individuals and the research objectives.
  Interventions: Behavioral: Tidal Model improvement model
- Tidal Model Control Group (No Intervention): Individuals in the control group will continue their lives.

INTERVENTIONS:
Behavioral: Tidal Model improvement model — 1. st interview Pre-assessment Application of measurement tools
  2. nd meeting Orientation Concept of recovery, change phase of the individual, Holistic Evaluation, Creation of Personal Safety Plan 3. Interview Process planning Setting goals, Starting One-on-One Sessions
  4th meeting Healing is possible, accepting his illness, overcoming change, emphasizing his strengths, instilling hope 5.-6. interview Empowerment Coping with crisis, reducing anxiety, relaxation exercises, individual roles, assertiveness, strengthening self-esteem 7.-8. Interview Maintaining control of life, taking responsibility for behavior, appropriate expression of anger, feeling, thinking and Taking responsibility for recovery, discovering behaviors 9th interview Creating a supportive environment Increasing new interactions, relationships, social skills 10th meeting Evaluation Finalizing the personal security plan, using new knowledge and behaviors in the healing journey, evaluation of the process
  Arms: Tidal Model improvement model

SUMMARY:
Aim:

In this study, it was aimed to evaluate the effect of the tidal model on distress, self-management and psychological well-being in individuals with diabetes. It is thought that this study will contribute to the literature, nursing profession and patients with diabetes.

DETAILED DESCRIPTION:
Population of the Research: The population of the research will be individuals who applied to Osmaniye State Hospital and were diagnosed with Diabetes at least 6 months ago. The sample of the research: The sample of the research is; In calculating the number of samples, the study of Savaşan and Çam named 'The Effect of the Psychiatric Nursing Approach Based on the Tidal Model on Coping and Self-esteem in People with Alcohol Dependency: A Randomized Trial' was taken as reference.At the end of the Tidal Model application, the effect size was calculated as 0.652 based on the difference between the self-esteem scores. In this context; A power of 0.80 and a margin of error of 0.05 for type 1 were taken, and it was deemed appropriate to take a total of 60 individuals, with a sample size of 30 individuals in the intervention and control groups. Sample size is based on independent t-test. It was decided to include more than 20% of the sample number calculated in terms of losses during the implementation of the study and statistical analysis. Accordingly, 36 intervention and 36 control groups will beResearch data

Literature-based Personal Information Form will be collected using Diabetes Distress Scale Type 2 Diabetes Self-Management Scale Psychological Well-Being Scale. In order to conduct the study, the approval of the Clinical Research Ethics Committee, written permission from the institution and written permission from the participants were obtained.In the study, in which the psychiatric nursing approach based on the Tidal Model is applied, approximately 6 and 10 individual interviews will be held with the individuals in the experimental group in addition to the routine treatment and follow-up in the Osmaniye State Hospital training hall. The control group will continue to receive routine treatment and follow-up. In order to provide individualized care to the individuals in the experimental group, initiatives will be implemented by starting individual interviews and in line with the goals of the individuals and the objectives of the research. Considering the basic processes of the Tidal Model, stages of care, basic approach and Tidal competencies, an interview plan including the details of the interviews with diabetes patients will be created and a meeting plan will be made with One-to-One Sessions. It will be concluded with an average of 6 and 10 interviews, depending on the situation of the individuals. tried to be formed. The number of samples was calculated in the G*Power 3.1 program.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with diabetes for at least 6 months, Individuals aged 18 and over will be included in the study.

Exclusion Criteria:

Patients with any psychiatric or neurological disorder that would prevent adequate communication will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
1. The effect of using the tidal model on the distress status of individuals with diabetes will be evaluated. | up to 6-10 weeks
  The DDS is a 17-item psychological measurement tool that uses a Likert scale with each item scored from 1 (no distress) to 6 (serious distress) to reflect distress experienced over the last month. The total score is calculated by dividing the sum of the answers by 17. A score of ≥3 is defined as T2DM-related distress. There are four subscales and subscale scores are also calculated by dividing the sum of subscale answers to the total question count of the subscale. Subscales are as follows: the emotional burden subscale with 5 questions, the physician-related distress subscale with 4 questions, the regimen-related distress subscale with 5 questions, and the interpersonal distress subscale with 3 questions.
The effect of using the tidal model on the self-management status of individuals with diabetes will be evaluated. | up to 6-10 weeks
  There are 8 items in the original scale of the Diabetes Self-Management Perception Scale. High participation in these items indicates low self-efficacy. For this reason, the 3 items mentioned were reverse scored compared to the other items. The lowest score that can be obtained from the scale is 7, and the highest score is 35. A high total score indicates that the individual has good awareness of diabetes management
The effect of using the tidal model on the psychological well-being of individuals with diabetes will be evaluated. | up to 6-10 weeks
  The scale is an 8-item 7-point Likert-type (1=totally disagree, 7=totally agree) self-assessment scale. High scores indicate higher psychological well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Ejdane Coşkun, Principal Investigator — Korkut Ata University Osmaniye, Center, Türkiye, 80000; Ayşe İNEL MANAV, Principal Investigator — Korkut Ata University Osmaniye, Center, Türkiye, 80000; Derya Atik, Principal Investigator — Korkut Ata University Osmaniye, Center, Türkiye, 80000
Locations (1):
- Türkiye, Osmaniye, Korkut Ata University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Don't share